CLINICAL TRIAL: NCT03270748
Title: Post Transplant High-Dose Cyclophosphamide as GvHD Prophylaxis in Patients Receiving 1-Antigen/Allele HLA Mismatched (7/8 Matched) Unrelated Hemopoietic Stem Cell Transplantation for Myeloid Malignancies
Brief Title: Post Transplant High-Dose Cy as GvHD Prophylaxis in 1 HLA Mismatched Unrelated HSCT for Myeloid Malignancies
Acronym: GITMO-PHYLOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GITMO-PHYLOS
Record Dates: First submitted 2017-08-24; First posted 2017-09-01 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Myeloid Malignancies
Keywords: Allogeneic hematopoietic stem cell transplantation; acute graft-versus-host disease; Unrelated donors; Post-transplant cyclophosphamide; Myeloid Malignancies; unrelated hematopoietic cell transplantation; GITMO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Experimental: Experimental The experimental consists in the application of a therapeutic strategy: post Transplant High-Dose Cyclophosphamide as GvHD Prophylaxis in Patients Receiving 1-Antigen/Allele HLA Mismatched (7/8 matched) Unrelated Hemopoietic Stem Cell Transplantation for Myeloid Malignancies Therapeutic intervention, namely conditioning regimen and GVHD prophylaxis, are based on standard current regimens: Busulfan 0,8 mg/kg 4 times per day during 2 h infusions for 4 consecutive days (from day -6 through day -3) Fludarabine 40 mg/m2 per day for 4 days (from day -6 through day -3); GvHD prophylaxis: Cyclosporine or Tacrolimus beginning day+5 up to at least 100 days. Micofenolate 15mg/kg twice a day from day +5 to +35.
  Interventions: Drug: GvHD prophylaxis

INTERVENTIONS:
Drug: GvHD prophylaxis — Cyclophosphamide 50 mg/kg intravenously day+3 and +4 (total dose:100 mg/kg).

SUMMARY:
The experimental treatment consists in the application of a therapeutic strategy with post Transplant High-Dose Cyclophosphamide as GvHD Prophylaxis in Patients Receiving 1-Antigen/Allele HLA Mismatched (7/8 matched) Unrelated Hemopoietic Stem Cell Transplantation for Myeloid Malignancies.

DETAILED DESCRIPTION:
The experimental treatment consists in the application of a therapeutic strategy with post Transplant High-Dose Cyclophosphamide as GvHD Prophylaxis in Patients Receiving 1-Antigen/Allele HLA Mismatched (7/8 matched) Unrelated Hemopoietic Stem Cell Transplantation for Myeloid Malignancies Allogeneic hematopoietic stem cell transplantation is a potentially curative therapy for a variety of hematologic malignancies due to two separate components: chemo/radiotherapy administered before the transplant (conditioning regimen) and the presence of immunocompetent cells in the graft, capable of inducing a "graft-versus-malignancy effect" also known as "GvL" effect. However, this immune-reaction usually carries the risk of detrimental effects seen as a multi-organ syndrome known as graft-versus-host disease (GvHD), which remains the most feared complication of Allogeneic hematopoietic stem cell transplantation. GvHD may be given to disparities between donor and recipient in presence of gene mismatches in the Major Histocompatibility Complex, also known as Human Leucocyte Antigen (HLA) system, or in any minor histocompatibility antigen. Thus, GvHD is obviously more common (and possibly more severe) in patients transplanted from HLA-mismatched donors as compared with those receiving grafts from HLA-matched donors.

A major limitation of allo-HSCT is the availability of a donor given that only a small percentage of patients has a HLA identical family donor. For the majority of patients (approximately 70%) who lack a HLA-identical sibling, alternative donors include HLA-matched unrelated donors and cord blood units. The chance of identifying a suitable marrow unrelated donor (MUD) in the international voluntary donor registries is limited by the frequency of a certain HLA genotype in the general population.

One of the alternative options in such cases is the use of a HLA-mismatched unrelated donor (MMUD). HLA-mismatching is defined as the presence of unshared antigens/alleles in recipient-donor pairs for HLA-A, -B, -C or DRB1 loci.

Patients undergoing MUD or MMUD transplants usually receive an intensified three-drug immunosuppressive regimen: anti-thymocyte globulin in addition to the standard platform of a calcineurine-inhibitor and an anti-metabolite.

The effect of HLA mismatches on clinical outcomes has been investigated in several studies. Single HLA mismatches at HLA-A, -B, -C, or -DRB1 locus (7/8 HLA-matched) were associated with lower overall survival and disease free survival, higher non-relapse mortality, and higher incidence of acute GvHD as compared with 8/8 HLA-matched pairs.

Many clinical trials suggest that high-dose Cy administrated after allogeneic HSCT didn't cause prolonged aplasia due toxicity on donor stem cells; could prevent rejection due to HLA-disparity and could be effective in preventing GvHD, allowing adequate immune-reconstitution.

With this study the investigators plan to investigate if post-transplant high-dose Cy, with a calcineurine inhibitor and mycophenolate, could reduce acute GvHD rates and infectious complications improving clinical outcomes of MMUD transplants in patients with acute myeloid leukemia and myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

Acute myeloid leukemia in complete remission Myelodysplastic syndrome Indication for allo-HCT No available HLA identical sibling donor or HLA matched unrelated donor Activation of an alternative donor search Presence of a 1 antigen/allele mismatched (7/8 HLA matched) unrelated donor ECOG performance status <2 Written and signed informed consent

Exclusion Criteria:

left ventricular ejection fraction < 40% FEV1, FVC, DLCO <50% of predicted LFT > 5 times the upper limit of normal creatinine clearance < 40 ml/min Previous allogeneic Hemopoietic Stem Cell Transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
incidence of acute GvHD | day +100 post-transplant
  cumulative incidence of acute GvHD (grade II-IV) at 100 days post Unrelated Hemopoietic Stem Cell Transplantation

SECONDARY OUTCOMES:
Overall survival | 1 year post transplantation
  is defined as the time from transplant to the date of death due to any cause or to the last date the patient was known to be alive (censored observation) or to the date of the data cut-off for final analysis
GRFS (GvHD free, relapse free survival) | first 12 months after transplantation
  are defined as occurrence of grade III-IV acute GvHD, chronic GvHD requiring systemic immunosuppressive treatment, disease relapse, or death from any cause
chronic graft-versus-host disease | 3 years from transplantation
  Cumulative incidence and severity of chronic graft-versus-host disease (by NIH criteria)
Graft failure | day +100 and 1 year after transplantation
  failure a) Primary graft failure is defined as < 5% donor chimerism. Secondary graft failure (graft rejection) is defined as initial recovery followed by neutropenia with <5% donor chimerism. b) Rate of graft rejection and graft failure
Haematopoietic Recovery | participants will be followed for the duration of hospital stay, an expected average of 30 days
  Time to reach an absolute neutrophil count > 0.5 109/L from day of HSCT. Neutrophil recovery end-point will be defined as the first of 3 consecutive days with an absolute neutrophil count > 0.5 x109/L. Time to reach platelet engraftment, defined as the number of days after HSCT (Day 0) for patients to maintain an un-transfused platelet count of > 20.0 x 109/L.
Non Relapse Mortality | at 100 days, at 180days and at 1 year from transplantation
  The cumulative incidence of Non Relapse Mortality is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation. Cumulative incidence
Relapse and Residual Disease | at 1 year from transplantation
  Testing for recurrent malignancy in the blood, marrow or other sites will be used to assess relapse after transplantation. For the purpose of this study, relapse is defined by either morphological or cytogenetic evidence of acute myeloid leukemia or myelodisplastic syndrome consistent with pre-transplant features. Molecular relapse will be defined where available as any evidence of a pre-transplant defined abnormality using conventional cytogenetics or FISH techniques or cytofluorimetric analysis or molecular probes
Incidence of infectious complications and kinetics of immune-reconstitution | one year after transplant
  the rate of proven and probable invasive fungal infections and viral reactivation/disease (CMV, HHV6,Adenovirus, EBV). Immune-reconstitution will be evaluated with lymphocyte sub-populations counts (CD3+, CD4+, CD8+, CD16+, CD20+) and IgG, IgA, IgM titer

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Raiola, MD, Principal Investigator — Ospedale Policlinico San Martino-IST
Locations (33):
- Italy (33):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Ospedali Riuniti, Ancona
  - Ospedale Moscati, Avellino
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale San Orsola, Bologna
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - ASST Spedali Civili, Brescia
  - Ospedale Binaghi, Cagliari
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - AOU-IRCCS San Martino-IST, Genova
  - Osp. Card. Panico, Lecce
  - AOU Integrata, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Niguarda Ca' Grande, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - ASST Ospedale S. Gerardo de' i Tintori - Università degli Studi di Milano, Monza
  - A.O.U. Policlinico Federico II, Napoli
  - Azienda ospedaliera Universitaria di Parma, Parma
  - Fondazione IRCCS San Matteo, Pavia
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - A.O. San Camillo Forlanini, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Az. Ospedaliera Universitaria Senese - Divisione Ematologia e Trapianti, Siena
  - Ospedale Moscati, Taranto
  - A.O.U. Citta della Salute e della Scienza, Torino
  - Ospedale Gonzaga, Torino
  - A.O. Santa Maria della Misericordia, Udine
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza

REFERENCES:
- [Derived] Raiola AM, Bruno B, Risitano AM, Mosna F, Cavattoni IM, Onida F, Saporiti G, Patriarca F, Battista ML, Pavone V, Mele A, Chiusolo P, Sica S, Loteta B, di Grazia C, Carella AM, Salvatore D, Morello E, Leoni A, Giaccone L, Bernasconi P, Terruzzi E, Mordini N, Borghero C, Zallio F, Luppi M, Grassi A, Olivieri A, Piras E, Sacchi N, Ciccone G, Castiglione A, Degrandi E, Angelucci E, Martino M, Bonifazi F. Posttransplant cyclophosphamide as GVHD prophylaxis in patients receiving mismatched unrelated HCT: the PHYLOS trial. Blood Adv. 2025 Apr 22;9(8):1966-1975. doi: 10.1182/bloodadvances.2024015173. PMID 39928954